CLINICAL TRIAL: NCT05920031
Title: Combining Cross-Education and Mirror Therapy for Upper Limb Rehabilitation in Post-Stroke Patients: A Randomized Controlled Trial
Brief Title: Cross-Education and Mirror Therapy for Upper Limb in Post-Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/0585850002023
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cross-education training only (Experimental): Participants will perform resistance exercises at 60% of their 1 repetition maximum (1RM) with the less affected limb.
  Interventions: Other: Cross-education
- Mirror therapy only (Experimental): Participants will perform bilateral upper limb movements while observing the reflection of the less affected limb in a mirror.
  Interventions: Other: Mirror therapy
- Combined cross-education and mirror therapy (Experimental): Participants will perform resistance exercises with the less affected limb while observing its reflection in a mirror.
  Interventions: Other: Cross-education; Other: Mirror therapy
- Conventional rehabilitation (Active Comparator): Participants will receive conventional rehabilitation for post-stroke upper limb motor impairments.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Cross-education — Participants will perform resistance exercises at 60% of their 1 repetition maximum (1RM) with the less affected limb. The intervention will be performed three times per week for 8 weeks. Each session will consist of three sets of 15 repetitions of bicep curls, tricep extensions, and wrist flexion/extension exercises with a 1-minute rest period between sets. The exercises will be performed in a seated position, with the participant's forearm resting on a table and the therapist providing manual resistance. The therapist will be positioned in front of the participant.
  Arms: Combined cross-education and mirror therapy; Cross-education training only
Other: Mirror therapy — Participants will perform bilateral upper limb movements while observing the reflection of the less affected limb in a mirror. The intervention will be performed three times per week for 8 weeks. Each session will consist of 10 minutes of mirror therapy, with the participant seated in front of a mirror. The participant will perform various upper limb movements, such as reaching and grasping, while observing the mirror reflection of the less affected limb. The therapist will be positioned beside the participant, providing verbal cues and feedback as necessary.
  Arms: Combined cross-education and mirror therapy; Mirror therapy only
Other: Conventional Physical Therapy — articipants will receive conventional rehabilitation for post-stroke upper limb motor impairments, which may include exercises such as range of motion, stretching, and strengthening of the affected limb, as well as other therapies such as electrical stimulation or constraint-induced movement therapy. The intervention will be individualized for each participant and will be performed three times per week for 8 weeks. The frequency, duration, and intensity of the exercises will be gradually increased over the course of the intervention, based on the participant's progress. The exercises may be performed in a seated or standing position, depending on the participant's ability and preference. The therapist will be positioned in front of or beside the participant, providing verbal cues and feedback as necessary.
  Arms: Conventional rehabilitation

SUMMARY:
This randomized controlled trial will investigate the potential synergistic effects of combining cross-education training with mirror therapy on strength and motor function in the more affected upper limb of post-stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Post-stroke patients with upper limb motor impairments
* Aged 30 years to 60 years old
* At least 3 months post-stroke
* Able to participate in the intervention

Exclusion Criteria:

* Severe cognitive impairments
* Visual impairments
* Any contraindications to the intervention

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-28 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Changes in Upper limb strength | Changes in Upper limb strength at baseline, 8 weeks, 16 weeks
  Upper limb strength (measured by hand-held dynamometry)
Changes in motor function | Changes in motor function at baseline, 8 weeks, 16 weeks
  motor function (measured by Fugl-Meyer Assessment)

SECONDARY OUTCOMES:
Changes in Quality of life | Changes in Quality of life at baseline, 8 weeks, 16 weeks
  Quality of life (measured by Stroke Impact Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No